CLINICAL TRIAL: NCT02949934
Title: Effects of Cortical Dopamine Regulation on Drinking, Craving, and Cognitive Control
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Raymond F. Anton, Distinguished University Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00050157; P50AA010761 (NIH)
Record Dates: First submitted 2016-10-26; First posted 2016-10-31 (Estimated); Results first posted 2022-04-15 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Tolcapone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo/rs4680 val/val (Placebo Comparator): Placebo three times per day for eight days
  Individuals with the rs4680 val/val genotype
  Interventions: Drug: Placebo
- Tolcapone/rs4680 val/val (Active Comparator): Tolcapone 100 mg three times per day for three days Tolcapone 200 mg three times per day for five days
  Individuals with the rs4680 val/val genotype
  Interventions: Drug: Tolcapone
- Placebo/rs4680 val/met (Placebo Comparator): Placebo three times per day for eight days
  Individuals with the rs4680 val/met genotype
  Interventions: Drug: Placebo
- Tolcapone/rs4680 val/met (Active Comparator): Tolcapone 100 mg three times per day for three days Tolcapone 200 mg three times per day for five days
  Individuals with the rs4680 val/met genotype
  Interventions: Drug: Tolcapone
- Placebo/rs4680 met/met (Placebo Comparator): Placebo three times per day for eight days
  Individuals with the rs4680 met/met genotype
  Interventions: Drug: Placebo
- Tolcapone/rs4680 met/met (Active Comparator): Tolcapone 100 mg three times per day for three days Tolcapone 200 mg three times per day for five days
  Individuals with the rs4680 met/met genotype
  Interventions: Drug: Tolcapone

INTERVENTIONS:
Drug: Tolcapone
  Other Names: Tasmar
  Arms: Tolcapone/rs4680 met/met; Tolcapone/rs4680 val/met; Tolcapone/rs4680 val/val
Drug: Placebo
  Arms: Placebo/rs4680 met/met; Placebo/rs4680 val/met; Placebo/rs4680 val/val

SUMMARY:
The purpose of this study is to determine whether the catechol-O-methyltransferase (COMT) inhibitor tolcapone, relative to placebo, reduces alcohol drinking and alcohol cue-elicited brain activation and increases brain activation associated with cognitive control as a function of a participant's genotype at a polymorphism in the COMT gene.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-40 (to focus on an age group still on a trajectory of increasing alcohol consumption).
2. Meets Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) criteria for current Alcohol Use Disorder.
3. Currently not engaged in, and does not want treatment for, alcohol-related problems.
4. Able to read and understand questionnaires and informed consent.
5. Lives within 50 miles of the study site.
6. Able to maintain abstinence from alcohol for two days (without the aid of detoxification medications), as determined by self report and breathalyzer measurements.

Exclusion Criteria:

1. Current DSM-5 diagnosis of any other substance use disorder except Nicotine Use Disorder.
2. Any psychoactive substance use (except marijuana and nicotine) within the last 30 days, as indicated by self-report and urine drug screen. For marijuana, no use within the last seven days by verbal report and negative (or decreasing) urine tetrahydrocannibinol (THC) levels.
3. Current DSM-5 Axis I diagnosis, including major depression, panic disorder, obsessive-compulsive disorder, post-traumatic stress disorder, bipolar affective disorder, schizophrenia, dissociative disorders, eating disorders, or any other psychotic or organic mental disorder.
4. Current suicidal ideation or homicidal ideation.
5. Need for maintenance or acute treatment with any psychoactive medication, including antiepileptic medications.
6. Currently taking medication known to affect alcohol intake (e.g., disulfiram, naltrexone, acamprosate, topiramate).
7. History of severe alcohol withdrawal (e.g., seizure, delirium tremens), as evidenced by self-report and assessment with Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA-Ar).
8. Clinically significant medical problems such as cardiovascular, renal, gastrointestinal, or endocrine problems that would impair participation or limit medication ingestion.
9. Past alcohol-related medical illness, such as gastrointestinal bleeding, pancreatitis, or peptic ulcer.
10. Current or past hepatocellular disease, as indicated by verbal report or elevations of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than the upper limit of the normal range at screening.
11. Females of childbearing potential who are pregnant (by urine human chorionic gonadotropin), nursing, or who are not using a reliable form of birth control.
12. Current charges pending for a violent crime (not including drinking while intoxicated).
13. Lack of a stable living situation.
14. Presence of ferrous metal in the body, as evidenced by metal screening and self-report.
15. Severe claustrophobia or morbid obesity that preclude placement in the MRI scanner.
16. History of head injury with > 2 minutes of unconsciousness.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-04-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schacht JP, Yeongbin Im, Hoffman M, Voronin KE, Book SW, Anton RF. Effects of pharmacological and genetic regulation of COMT activity in alcohol use disorder: a randomized, placebo-controlled trial of tolcapone. Neuropsychopharmacology. 2022 Oct;47(11):1953-1960. doi: 10.1038/s41386-022-01335-z. Epub 2022 May 6. PMID 35523943

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were genotyped for the COMT rs4680 single nucleotide polymorphism and subsequently randomized, on the basis of their rs4680 genotype, to take tolcapone or placebo for eight days. Outcomes were the number of standard alcoholic drinks consumed during Days 1-6 ("Natural Drinking Period"), alcohol cue-elicited brain activation on Day 7 ("Neuroimaging"), and the number of drinks, out of 8 possible, that participants chose to self-administer in the lab on Day 8 ("Bar Laboratory").
Period: Natural Drinking Period
Arm/Group | Placebo/rs4680 Val/Val | Tolcapone/rs4680 Val/Val | Placebo/rs4680 Val/Met | Tolcapone/rs4680 Val/Met | Placebo/rs4680 Met/Met | Tolcapone/rs4680 Met/Met
Started | 16 | 12 | 17 | 16 | 15 | 14
Completed | 15 | 12 | 17 | 15 | 14 | 14
Not Completed | 1 | 0 | 0 | 1 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0
Period: Neuroimaging
Arm/Group | Placebo/rs4680 Val/Val | Tolcapone/rs4680 Val/Val | Placebo/rs4680 Val/Met | Tolcapone/rs4680 Val/Met | Placebo/rs4680 Met/Met | Tolcapone/rs4680 Met/Met
Started | 15 | 12 | 17 | 15 | 14 | 14
Completed | 12 | 12 | 15 | 15 | 12 | 12
Not Completed | 3 | 0 | 2 | 0 | 2 | 2
Not completed — Protocol Violation | 2 | 0 | 0 | 0 | 1 | 0
Not completed — Motion artifacts in imaging data | 1 | 0 | 1 | 0 | 1 | 0
Not completed — Not scanned | 0 | 0 | 1 | 0 | 0 | 2
Period: Bar Laboratory
Arm/Group | Placebo/rs4680 Val/Val | Tolcapone/rs4680 Val/Val | Placebo/rs4680 Val/Met | Tolcapone/rs4680 Val/Met | Placebo/rs4680 Met/Met | Tolcapone/rs4680 Met/Met
Started (The number of participants who started the bar laboratory on Day 8 is in some cases greater than the number who completed neuroimaging on Day 7. Some participants were not scanned on Day 7 and some had unusable neuroimaging data due to motion, but still started the bar laboratory.) | 13 | 12 | 17 | 15 | 13 | 14
Completed | 12 | 7 | 10 | 11 | 7 | 13
Not Completed | 1 | 5 | 7 | 4 | 6 | 1
Not completed — Procedure not done due to COVID-19 pandemic | 0 | 5 | 5 | 3 | 5 | 1
Not completed — Adverse Event | 1 | 0 | 2 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Non-treatment-seeking individuals between the ages of 21 and 40 with DSM-5 diagnosed Alcohol Use Disorder.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/rs4680 Val/Val | Tolcapone/rs4680 Val/Val | Placebo/rs4680 Val/Met | Tolcapone/rs4680 Val/Met | Placebo/rs4680 Met/Met | Tolcapone/rs4680 Met/Met | Total
Number analyzed (Participants) | 16 | 12 | 17 | 16 | 15 | 14 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.9 (5.5) | 29.3 (4.7) | 25.7 (4.7) | 26.3 (5.0) | 26.3 (5.2) | 25.3 (5.7) | 26.5 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 5 | 6 | 6 | 9 | 37
  Male | 11 | 6 | 12 | 10 | 9 | 5 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 1 | 0 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 2 | 1 | 0 | 1 | 7
  White | 12 | 11 | 15 | 14 | 15 | 12 | 79
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 12 | 17 | 16 | 15 | 14 | 90

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Standard Drinks Per Day Consumed During Natural (Usual Environment) Conditions
Description: Number of standard alcoholic drinks per day that participants reported consuming, as assessed by the Timeline Follow-back method.
Time Frame: Days 1-6 of study medication ingestion
Measure: Mean (Standard Error); unit: standard drinks per day
Arm/Group | Placebo/rs4680 Val/Val | Tolcapone/rs4680 Val/Val | Placebo/rs4680 Val/Met | Tolcapone/rs4680 Val/Met | Placebo/rs4680 Met/Met | Tolcapone/rs4680 Met/Met
Number analyzed (Participants) | 15 | 12 | 17 | 15 | 14 | 14
standard drinks per day | 6.018 (0.586) | 3.534 (0.668) | 3.998 (0.538) | 5.012 (0.567) | 5.271 (0.596) | 5.949 (0.602)
Statistical Analysis 1: Comparison: Placebo/rs4680 Val/Val vs Tolcapone/rs4680 Val/Val vs Placebo/rs4680 Val/Met vs Tolcapone/rs4680 Val/Met vs Placebo/rs4680 Met/Met vs Tolcapone/rs4680 Met/Met; Analysis was an ANCOVA testing the interaction between rs4680 genotype and medication group; Test type: Superiority; p = 0.013, ANCOVA; Covariates were age, baseline AUDIT score, baseline drinks per day, and whether participant participated before vs. during the COVID-19 pandemic

2. Primary Outcome: Total Number of Drinks Under Controlled Conditions (Bar Lab)
Description: Total number of drinks, out of 8 possible, that participants chose to consume in the bar laboratory after receipt of a priming drink, targeted by sex and body weight to produce a breath alcohol concentration of 0.03 g/dL. Each of the drinks that participants chose to consume was targeted to produce a breath alcohol concentration of 0.015 g/dL. Participants were given a "bar credit" of $16 with which to "purchase" drinks, at the cost of $2/drink, and were told that any money they did not spend would be given to them the following day.
Time Frame: 2 hours during the alcohol challenge procedure
Population: Due to the COVID-19 pandemic and the need for social distancing, a protocol amendment was required to remove the bar lab procedure. Thus, this outcome was assessed for only the first 63 participants.
Measure: Mean (Standard Error); unit: Drinks
Arm/Group | Placebo/rs4680 Val/Val | Tolcapone/rs4680 Val/Val | Placebo/rs4680 Val/Met | Tolcapone/rs4680 Val/Met | Placebo/rs4680 Met/Met | Tolcapone/rs4680 Met/Met
Number analyzed (Participants) | 14 | 7 | 10 | 11 | 8 | 13
Drinks | 5.353 (0.721) | 3.256 (0.955) | 5.01 (0.812) | 4.964 (0.752) | 1.68 (0.935) | 4.732 (0.704)
Statistical Analysis 1: Comparison: Placebo/rs4680 Val/Val vs Tolcapone/rs4680 Val/Val vs Placebo/rs4680 Val/Met vs Tolcapone/rs4680 Val/Met vs Placebo/rs4680 Met/Met vs Tolcapone/rs4680 Met/Met; Analysis was an ANCOVA testing the interaction between rs4680 genotype and medication group; Test type: Superiority; p = 0.014, ANCOVA; Covariates were age, baseline AUDIT score, and baseline drinks per day

3. Other Pre Specified Outcome: Cognitive-control-associated Brain Activation (fMRI)
Description: Magnitude of change between baseline and day 7 scan in the BOLD signal in the right inferior frontal gyrus to spatial working memory
Time Frame: 7 days--change between baseline and scan on day 7
Population: Participants who completed both fMRI scans and had usable data
Measure: Mean (Standard Error); unit: Arbitrary units (Day 7 minus Baseline)
Groups:
- Placebo/rs4680 Val/Val: Placebo three times per day for eight days
  Individuals with the rs4680 val/val genotype
  Placebo
- Tolcapone/rs4680 Val/Val: Tolcapone 100 mg three times per day for three days Tolcapone 200 mg three times per day for five days
  Individuals with the rs4680 val/val genotype
  Tolcapone
- Placebo/rs4680 Val/Met: Placebo three times per day for eight days
  Individuals with the rs4680 val/met genotype
  Placebo
- Tolcapone/rs4680 Val/Met: Tolcapone 100 mg three times per day for three days Tolcapone 200 mg three times per day for five days
  Individuals with the rs4680 val/met genotype
  Tolcapone
- Placebo/rs4680 Met/Met: Placebo three times per day for eight days
  Individuals with the rs4680 met/met genotype
  Placebo
- Tolcapone/rs4680 Met/Met: Tolcapone 100 mg three times per day for three days Tolcapone 200 mg three times per day for five days
  Individuals with the rs4680 met/met genotype
  Tolcapone
Arm/Group | Placebo/rs4680 Val/Val | Tolcapone/rs4680 Val/Val | Placebo/rs4680 Val/Met | Tolcapone/rs4680 Val/Met | Placebo/rs4680 Met/Met | Tolcapone/rs4680 Met/Met
Number analyzed (Participants) | 11 | 12 | 15 | 14 | 12 | 11
Arbitrary units (Day 7 minus Baseline) | -0.196 (.086) | -0.063 (.082) | -0.178 (.074) | 0.076 (.076) | -0.017 (.082) | -0.224 (.086)
Statistical Analysis 1: Comparison: Placebo/rs4680 Val/Val vs Tolcapone/rs4680 Val/Val vs Placebo/rs4680 Val/Met vs Tolcapone/rs4680 Val/Met vs Placebo/rs4680 Met/Met vs Tolcapone/rs4680 Met/Met; Test type: Superiority; p = 0.062, Mixed Models Analysis; Linear mixed model testing interaction between rs4680 genotype, medication group, and time, controlling for scanner

4. Other Pre Specified Outcome: Alcohol Cue-elicited Brain Activation (fMRI)
Description: Magnitude of change between baseline and day 7 scan in the right inferior frontal gyrus blood oxygenation level dependent (BOLD) signal to alcohol cues, relative to neutral beverage cues (alcohol cue reactivity task described in Schacht et al., 2013, Neuropsychopharmacology)
Time Frame: 7 days--change between baseline and scan on day 7
Population: Participants who completed both fMRI scans and had usable scan data
Measure: Mean (Standard Error); unit: Arbitrary units (Day 7 minus Baseline)
Arm/Group | Placebo/rs4680 Val/Val | Tolcapone/rs4680 Val/Val | Placebo/rs4680 Val/Met | Tolcapone/rs4680 Val/Met | Placebo/rs4680 Met/Met | Tolcapone/rs4680 Met/Met
Number analyzed (Participants) | 12 | 12 | 15 | 15 | 12 | 12
Arbitrary units (Day 7 minus Baseline) | 0.09 (.070) | -0.045 (.070) | 0.066 (.063) | -0.164 (.063) | 0.138 (.070) | .006 (.070)
Statistical Analysis 1: Comparison: Placebo/rs4680 Val/Val vs Tolcapone/rs4680 Val/Val vs Placebo/rs4680 Val/Met vs Tolcapone/rs4680 Val/Met vs Placebo/rs4680 Met/Met vs Tolcapone/rs4680 Met/Met; Test type: Superiority; p = 0.83, Mixed Models Analysis; Linear mixed model testing interaction between rs4680 genotype, medication group, and time, controlling for scanner
Statistical Analysis 2: Comparison: Placebo/rs4680 Val/Val vs Tolcapone/rs4680 Val/Val vs Placebo/rs4680 Val/Met vs Tolcapone/rs4680 Val/Met vs Placebo/rs4680 Met/Met vs Tolcapone/rs4680 Met/Met; Test type: Superiority; p = 0.026, Mixed Models Analysis; Linear mixed model testing interaction between medication group and time, controlling for scanner

ADVERSE EVENTS:
Time Frame: 8 days
Arm/Group | Placebo/rs4680 Val/Val | Tolcapone/rs4680 Val/Val | Placebo/rs4680 Val/Met | Tolcapone/rs4680 Val/Met | Placebo/rs4680 Met/Met | Tolcapone/rs4680 Met/Met
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/12 | 0/17 | 0/16 | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/12 | 0/17 | 0/16 | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 1/16 | 0/12 | 0/17 | 1/16 | 0/15 | 0/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/rs4680 Val/Val (N=16) | Tolcapone/rs4680 Val/Val (N=12) | Placebo/rs4680 Val/Met (N=17) | Tolcapone/rs4680 Val/Met (N=16) | Placebo/rs4680 Met/Met (N=15) | Tolcapone/rs4680 Met/Met (N=14)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-11): https://cdn.clinicaltrials.gov/large-docs/34/NCT02949934/Prot_SAP_000.pdf